CLINICAL TRIAL: NCT01309997
Title: A Randomized Phase II Study of Imatinib and Rituximab for Cutaneous Sclerosis After Allogeneic Hematopoietic Cell Transplantation
Brief Title: Imatinib and Rituximab in Treating Cutaneous Sclerosis in Patients With Chronic Graft-Versus-Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lee, Stephanie (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Lee, Stephanie, Principal Investigator, Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Organization: Fred Hutchinson Cancer Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2343.00; NCI-2011-00098 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RDCRN 6502 (Other: Rare Diseases Clinical Research Network II); 2343.00 (Other: Fred Hutchinson Cancer Research Center); U54CA163438 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2011-03-01; First posted 2011-03-07 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-05

CONDITIONS: Graft Versus Host Disease; Systemic Scleroderma
Keywords: Imatinib; Rituximab; Chronic Graft-vs-Host Disease
MeSH Terms: conditions — Graft vs Host Disease; Scleroderma, Systemic | interventions — Imatinib Mesylate; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (enzyme inhibitor) (Experimental): Patients receive imatinib mesylate PO QD for 6 months in the absence of progression of sclerosis or unacceptable toxicity.
  Interventions: Drug: imatinib mesylate
- Arm II (monoclonal antibody) (Experimental): Patients receive rituximab IV on days 1, 8, 15, and 22. A second treatment cycle is repeated at 3 months for a total of 8 doses of rituximab in the absence of progression of sclerosis or unacceptable toxicity.
  Interventions: Biological: rituximab

INTERVENTIONS:
Drug: imatinib mesylate — Given PO
  Other Names: CGP 57148; Gleevec; Glivec
  Arms: Arm I (enzyme inhibitor)
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
  Arms: Arm II (monoclonal antibody)

SUMMARY:
This randomized phase II trial is evaluating how well imatinib mesylate works compared to rituximab in treating cutaneous sclerosis in patients with chronic graft- versus-host disease (GVHD). Both imatinib and rituximab have been reported to decrease skin thickening and improve skin and joint flexibility in people with cutaneous sclerosis due to chronic GVHD.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the best clinical response rate of cutaneous sclerosis (skin and/or fascial thickening) after 6 months of initial therapy with either imatinib (imatinib mesylate) or rituximab.

SECONDARY OBJECTIVES:

I. To determine the best response at either the 3 or 6 month assessment.

II. To determine the response rate at the 3 month assessment.

III. To determine the proportion of subjects who are able to taper corticosteroid after 6 months of imatinib or rituximab therapy.

IV. To determine the incidence of treatment failure to initial treatment with either imatinib or rituximab.

V. To evaluate if the Scleroderma Health Assessment Questionnaire (SHAQ) findings correlate with severity of cutaneous sclerosis clinical findings and response to study treatment.

VI. To correlate the detection of antibody against platelet derived growth factor receptor alpha (PDGFR A) with clinical response.

VII. To correlate change in B cell relevant parameters from baseline to 6 months or early crossover (antibody levels, skin collagen expression, B cell subsets) with therapeutic agent and best clinical response while on initial treatment.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive imatinib mesylate by mouth (PO) once daily (QD) for 6 months in the absence of progression of sclerosis or unacceptable toxicity. Subjects with a significant clinical response will continue to receive study drug for an additional 6 months.

ARM II: Patients receive rituximab intravenously (IV) on days 1, 8, 15, and 22 (first cycle). A second cycle of treatment with rituximab is repeated at 3 months for a total of 8 doses of rituximab in the absence of progression of sclerosis or unacceptable toxicity.

Patients with progression, treatment intolerance at any time up to 6 months, or no clinical response at 6 months will crossover to the other treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis within the past 18 months of cutaneous sclerosis after hematopoietic cell transplant (HCT) with sclerotic skin, morphea, myofascial involvement or joint contractures; must have a score of 2 or greater on the Vienna skin scale in any area, or a range-of-motion (ROM) score of 5 or less at the shoulder, elbow or wrist, or 3 or less at the ankle
* No medication added for the treatment of graft versus host disease (GVHD) within the past 4 weeks
* Receiving corticosteroids at a dose greater than required for treatment of adrenal insufficiency, unless the physician documents why steroids are contraindicated
* Age 2-99 years
* Karnofsky performance status >= 60% at enrollment
* All females of childbearing potential must have a negative serum or urine pregnancy test =< 7 days prior to starting study therapy
* All females of childbearing potential must agree to use a form of Food and Drug Administration (FDA) approved contraception from enrollment to one month after study treatment ends
* Subject has the ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Total bilirubin > 1.5x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 x ULN
* Renal insufficiency (serum creatinine > 2.0 mg/dl)
* Platelets < 30,000/ul or absolute neutrophil count < 1500/ul
* Known hypersensitivity to rituximab or other anti-B cell antibodies
* Known imatinib intolerance or allergy
* Evidence of any active viral, bacterial, or fungal infection that is progressive despite appropriate treatment
* Hepatitis B surface antigen positive
* Hepatitis B core antibody positive, unless hepatitis B virus (HBV) deoxyribonucleic acid (DNA) is undetectable
* Hepatitis C antibody positive, unless hepatitis C virus (HCV) ribonucleic acid (RNA) is undetectable
* Pregnant, lactating, or planning a pregnancy while in the study
* Distal leg skin score 3 or higher as the only manifestation of sclerosis
* Prior treatment of chronic GVHD with imatinib, rituximab, or any other monoclonal B-cell antibody (e.g. ofatumumab)
* Receipt of imatinib within the previous 6 months for any indication
* Receipt of any monoclonal B-cell antibody (e.g. rituximab, ofatumumab) within the previous 12 months for any indication
* Treatment with anti-B-cell cellular therapy (e.g. chimeric antigen-receptor-engineered cells) at any time after transplant
* Current treatment with extracorporeal photopheresis (ECP) at the time of enrollment
* History of psychiatric disorder that would interfere with normal participation in this study
* Inability or unwillingness of subject and/or parent guardian to provide informed consent or comply with study protocol
* Use of non-FDA approved drugs within 4 weeks of participation
* Patient with any condition that, in the opinion of the investigator, would interfere with the subject's ability to comply with the study requirements
* Patients with uncontrolled substance abuse

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-03; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lee, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (10):
- United States (10):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Stanford University Hospitals and Clinics, Stanford, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medical College, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient data and samples may be available with the appropriate approvals. Contact the PI for information.

REFERENCES:
- [Result] Arai S, Pidala J, Pusic I, Chai X, Jaglowski S, Khera N, Palmer J, Chen GL, Jagasia MH, Mayer SA, Wood WA, Green M, Hyun TS, Inamoto Y, Storer BE, Miklos DB, Shulman HM, Martin PJ, Sarantopoulos S, Lee SJ, Flowers ME. A Randomized Phase II Crossover Study of Imatinib or Rituximab for Cutaneous Sclerosis after Hematopoietic Cell Transplantation. Clin Cancer Res. 2016 Jan 15;22(2):319-27. doi: 10.1158/1078-0432.CCR-15-1443. Epub 2015 Sep 16. PMID 26378033

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Enzyme Inhibitor): Patients receive imatinib mesylate PO QD for 6 months in the absence of progression of sclerosis or unacceptable toxicity. During the 6mo study treatment period, if drug intolerance or disease progression is observed, they are crossed over to rituximab.
- Arm II (Monoclonal Antibody): Patients receive rituximab IV on days 1, 8, 15, and 22. A second treatment cycle is repeated at 3 months for a total of 8 doses of rituximab in the absence of progression of sclerosis or unacceptable toxicity. During the 6mo study treatment period, if drug intolerance or disease progression is observed, they are crossed over to imatinib.
Period: Overall Study
Arm/Group | Arm I (Enzyme Inhibitor) | Arm II (Monoclonal Antibody)
Started | 35 | 37
Remained on First Arm Only | 16 | 14
Crossed Over to Second Arm | 19 | 23
Completed | 30 | 31
Not Completed | 5 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 3
Not completed — Lack of Efficacy | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm II (Monoclonal Antibody): Patients receive rituximab IV on days 1, 8, 15, and 22. A second treatment cycle is repeated at 3 months for a total of 8 doses of rituximab in the absence of progression of sclerosis or unacceptable toxicity. TDuring the 6mo study treatment period, if drug intolerance or disease progression is observed, they are crossed over to imatinib.
- Total: Total of all reporting groups
Arm/Group | Arm I (Enzyme Inhibitor) | Arm II (Monoclonal Antibody) | Total
Number analyzed (Participants) | 35 | 37 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 30 | 61
  >=65 years | 4 | 7 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Significant Clinical Response
Description: Assessed by decline in an affected area's skin score as measured with the Vienna Skin Scale (from 4 [worst] to 2, 3 to 1, or 2 to 0 [best]) without a concurrent increase of two or more points in another area OR by an increase in the range of motion of the shoulders, elbows or wrists by two points (in a 1-7 scale where 1 is worst and 7 is best) or of the ankles by one point (in a 1 to 4 scale where 1 is worst and 4 is best) without a concurrent worsening in another area.
Time Frame: 6 months
Population: Patients were not eligible for evaluation if they discontinued participation or had missing 6 mo data.
Measure: Number; unit: participants
Groups:
- Arm I (Enzyme Inhibitor): Patients who were randomized to receive imatinib mesylate PO QD for 6 months in the absence of progression of sclerosis or unacceptable toxicity.
- Arm II (Monoclonal Antibody): Patients who were randomized to receive rituximab IV on days 1, 8, 15, and 22. A second treatment cycle was repeated at 3 months for a total of 8 doses of rituximab in the absence of progression of sclerosis or unacceptable toxicity.
Arm/Group | Arm I (Enzyme Inhibitor) | Arm II (Monoclonal Antibody)
Number analyzed (Participants) | 30 | 31
participants | 9 | 10

2. Secondary Outcome: Patients Who Were Able to Taper Corticosteroids
Description: Patients who achieved a greater than or equal to 50% reduction in the daily corticosteroid dose at 6mo compared to baseline
Time Frame: 6 months
Population: Patients with no corticosteroid dose data missing from baseline or 6mo.
Measure: Number; unit: participants
Groups:
- Arm I (Enzyme Inhibitor): Patients randomized to receive imatinib mesylate as their first therapy. They may take this from 1 mo-18 mo.
- Arm II (Monoclonal Antibody): Patients randomized to receive rituximab IV as their first therapy. They may receive from 1-2 four week cycles.
Arm/Group | Arm I (Enzyme Inhibitor) | Arm II (Monoclonal Antibody)
Number analyzed (Participants) | 27 | 32
participants | 7 | 9

3. Secondary Outcome: Cumulative Incidence of Treatment Failure
Description: Defined as discontinuation of randomized treatment due to chronic GVHD progression or treatment intolerance or no significant clinical response in sclerosis.
Time Frame: 6 months
Population: Only patients who were evaluable for SCR are included.
Measure: Number; unit: participants
Groups:
- Arm I (Enzyme Inhibitor): Patients randomized to receive imatinib mesylate PO QD as their first therapy. They may take this from 1 mo-18 mo.
Arm/Group | Arm I (Enzyme Inhibitor) | Arm II (Monoclonal Antibody)
Number analyzed (Participants) | 30 | 31
participants | 24 | 26

4. Secondary Outcome: Number of Patients Achieving Improvement in Cutaneous Sclerosis
Description: Assessed by decrease of >= 0.2 units (where 0 is best and 3.0 is worst ) in the Scleroderma Health Assessment Questionnaire (SHAQ).
Time Frame: 6 months
Population: Only patients evaluable at 6 mo are included.
Measure: Number; unit: participants
Groups:
- Arm 1 (Enzyme Inhibitor): Patients randomized to receive imatinib mesylate PO QD as their first therapy. They may take this from 1 mo-18 mo.
- Arm II (Monocolonal Antibody): Patients randomized to receive rituximab IV as their first therapy. They may receive from 1-2 four week cycles.
Arm/Group | Arm 1 (Enzyme Inhibitor) | Arm II (Monocolonal Antibody)
Number analyzed (Participants) | 30 | 31
participants | 2 | 9

5. Secondary Outcome: Baseline Histopathologic Score in the Two Treatment Arms
Description: Instrument: Nash dermal fibrosis grade. Measures extent of sclerosis in skin biopsies by histologic examination. Scale ranges from grade 0-5. Nash grade 5 is most severe fibrosis (0 is better outcome, 5 is worse outcome). No subscales are used in Nash grade. Please see table 1 in the reference for grading of dermal fibrosis.
  Nash RA, McSweeney PA, Crofford LJ, Abidi M, Chen CS, Godwin JD, et al. High-dose immunosuppressive therapy and autologous hematopoietic cell transplantation for severe systemic sclerosis: long-term follow-up of the US multicenter pilot study. Blood 2007;110:1388-96.
Time Frame: Enrollment
Population: Only patients with skin biopsies at enrollment are included.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Arm 1 (Enzyme Inhibitor) | Arm II (Monoclonal Antibody)
Number analyzed (Participants) | 32 | 31
units on a scale | 2 [0 to 5] | 2 [0 to 5]

6. Secondary Outcome: Patients With Any Percentage Decline in Any Grade of Sclerosis Without Increase in Percentage of Higher Grades of Sclerosis in Other Areas on the Vienna Skin Scale
Description: Maximum of 10 body areas. Each area can be graded 0 (best) to 4 (worst). Each of those grades requires a percentage of involvement. Improvement is measured by reduction of involvement in any grade and any body area.
Time Frame: 6 months
Population: Only patients who were evaluable at 6mo are included.
Measure: Number; unit: participants
Arm/Group | Arm I (Enzyme Inhibitor) | Arm II (Monoclonal Antibody)
Number analyzed (Participants) | 30 | 31
participants | 14 | 9

7. Secondary Outcome: Percentage of CD27+ B Cells in Responders (SCR) and Non-responders
Description: %CD27+ B cells
Time Frame: 6 months
Measure: Mean (Full Range); unit: percentage of CD27+ B cells
Groups:
- Rituximab Responders: Attained a SCR with rituximab
- Rituximab Non-responders: Did not attain a SCR with rituximab
- Imatinib Responders: Attained a SCR with imatinib
- Imatinib Nonresponders: Did not attain a SCR with imatinib
Arm/Group | Rituximab Responders | Rituximab Non-responders | Imatinib Responders | Imatinib Nonresponders
Number analyzed (Participants) | 3 | 10 | 3 | 11
percentage of CD27+ B cells | 10 [5 to 17] | 4.3 [0 to 9] | 14.2 [5.2 to 21.6] | 17.1 [4.8 to 23.7]
Statistical Analysis 1: Comparison: Rituximab Responders vs Rituximab Non-responders; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Imatinib Responders vs Imatinib Nonresponders; Test type: Superiority or Other; p = 0.64, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 18 months
Groups:
- Imatinib as Initial Therapy: Arm I = imatinib, adverse event occurred after the start date of imatinib and if applicable, prior to start date of rituximab.
- Rituximab as Initial Therapy: Arm I = rituximab, adverse event occurred after the start date of rituximab and if applicable, prior to start date of imatinib.
- Imatinib as Secondary Therapy: Arm II = imatinib, adverse event occurred after the start date of imatinib. (All participants in this group received rituximab prior).
- Rituximab as Secondary Therapy: Arm II = rituximab, adverse event occurred after the start date of rituximab. (All participants in this group received imatinib prior).
Arm/Group | Imatinib as Initial Therapy | Rituximab as Initial Therapy | Imatinib as Secondary Therapy | Rituximab as Secondary Therapy
Serious Adverse Events (participants affected / at risk) | 11/35 | 19/37 | 19/23 | 15/19
Other Adverse Events (participants affected / at risk) | 12/35 | 12/37 | 21/23 | 1/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib as Initial Therapy (N=35) | Rituximab as Initial Therapy (N=37) | Imatinib as Secondary Therapy (N=23) | Rituximab as Secondary Therapy (N=19)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
INR increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other, specify: congestive heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Other, specify: coronary vasculopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other, specify: Pneumoperitoneum (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 2 (3) | 4 (4) | 1 (1)
Other specify: Norovirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other, specify: unknown etiology (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Other, specify: mastectomy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Other, specify: brain tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib as Initial Therapy (N=35) | Rituximab as Initial Therapy (N=37) | Imatinib as Secondary Therapy (N=23) | Rituximab as Secondary Therapy (N=19)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (4) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Forced expiratory volume decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 3 (3) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 1 (1) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other, specify: squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No